CLINICAL TRIAL: NCT02409511
Title: Microalbuminuria as a Cardiovascular Risk Factor (PRECISED Substudy)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PRECISED Substudy
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2016-11

CONDITIONS: Microalbuminuria; Endothelial Dysfunction; Diabetic Nephropathy; Diabetic Retinopathy
Keywords: Type 1 Diabetic; Type 2 Diabetic; Hypertension; Renal Injury; Diabetic retinopathy
MeSH Terms: conditions — Diabetic Nephropathies; Diabetic Retinopathy; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Type 1 diabetic, retinopathy, non cardiovascular disease: Type 1 diabetic patients with microalbuminuria, diabetic retinopathy and without cardiovascular disease
  Interventions: Other: non intervention
- Non-diabetic, hipertension: Non-diabetic patients with hypertension and microalbuminuria
  Interventions: Other: non intervention
- Type 2 diabetic, non diabetic retinopathy: Type 2 diabetic patients without diabetic retinopathy and microalbuminuria
  Interventions: Other: non intervention
- Type 2 diabetic with diabetic retinopathy: Type 2 diabetic patients with diabetic retinopathy and microalbuminuria
  Interventions: Other: non intervention
- Type 2 diabetic, with proven nephropathy: Type 2 diabetic patients with biopsy proven diabetic nephropathy.
  Interventions: Other: non intervention

INTERVENTIONS:
Other: non intervention

SUMMARY:
Microalbuminuria (MA) is an independent cardiovascular risk factor in diabetic and non-diabetic subjects.

However, in the setting of type 2 diabetes, microalbuminuria could be a marker of either early diabetic nephropathy or diffuse endothelial dysfunction. At present, there are no biomarkers that permit us to discriminate between these two conditions.

DETAILED DESCRIPTION:
A hypothesis free approach by using proteomic/metabolomic analyses in the urine samples of selected populations seems an appropriate approach by which to explore this issue. In addition, a driven hypothesis in the same groups of patients based on a sensitive marker of kidney injury also seems appropriate.

Urinary levels of KIM-1(Kidney Injury Molecule-1 ) have been found elevated in experimental diabetic nephropathy even before that MA . In addition, urinary levels of KIM-1 were found significantly elevated in type 1 diabetic patients with MA, in comparison with diabetics with normoalbuminuria and non-diabetic healthy controls. Moreover, low urinary KIM-1 levels at baseline were associated with the regression of MA during a follow-up of 2 years . Therefore, it could be hypothesized that the presence of MA + KIM-1 in urine samples would indicate renal injury rather than endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with diabetes mellitus type 2 with microalbuminuria with and without retinopathy.

Control groups: diabetes mellitus type 1 with microalbuminuria and retinopathy hypertensive patients with microalbuminuria and diabetic patients with a renal biopsy

Exclusion Criteria:

* Patients without microalbuminuria or patients with macroalbuminuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with diabetes mellitus type 2 with microalbuminuria with and without retinopathy.
  Control groups: diabetes mellitus type 1 with microalbuminuria and retinopathy hypertensive patients with microalbuminuria and diabetic patients with a renal biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-09 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
To find markers for a better definition of the meaning of microalbuminuria | 3 years
  Improve diagnosis of diabetic nephropathy
Complementary markers for improving the performance of MA | 3 years
  Improve diagnosis of diabetic nephropathy

SECONDARY OUTCOMES:
To identify candidates which could help to discriminate whether microalbuminuria is related to endothelial dysfunction rather than kidney damage | 3 years
To test whether the enhancement of this specific marker of kidney injury is able to identify those patients in which MA really means diabetic nephropathy. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Han WK, Bailly V, Abichandani R, Thadhani R, Bonventre JV. Kidney Injury Molecule-1 (KIM-1): a novel biomarker for human renal proximal tubule injury. Kidney Int. 2002 Jul;62(1):237-44. doi: 10.1046/j.1523-1755.2002.00433.x. PMID 12081583
- [Background] Huo W, Zhang K, Nie Z, Li Q, Jin F. Kidney injury molecule-1 (KIM-1): a novel kidney-specific injury molecule playing potential double-edged functions in kidney injury. Transplant Rev (Orlando). 2010 Jul;24(3):143-6. doi: 10.1016/j.trre.2010.02.002. Epub 2010 May 6. PMID 20447817
- [Background] Alter ML, Kretschmer A, Von Websky K, Tsuprykov O, Reichetzeder C, Simon A, Stasch JP, Hocher B. Early urinary and plasma biomarkers for experimental diabetic nephropathy. Clin Lab. 2012;58(7-8):659-71. PMID 22997966
- [Background] Vaidya VS, Niewczas MA, Ficociello LH, Johnson AC, Collings FB, Warram JH, Krolewski AS, Bonventre JV. Regression of microalbuminuria in type 1 diabetes is associated with lower levels of urinary tubular injury biomarkers, kidney injury molecule-1, and N-acetyl-beta-D-glucosaminidase. Kidney Int. 2011 Feb;79(4):464-70. doi: 10.1038/ki.2010.404. Epub 2010 Oct 27. PMID 20980978